CLINICAL TRIAL: NCT07079813
Title: Clinical Study on the Efficiency of Rapid Arrhythmia Mapping Using EasyStars™ High Density Mapping Catheter Applications
Acronym: Rapid Arrhythm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNZGQ01
Record Dates: First submitted 2025-06-12; First posted 2025-07-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Tachycardia (VT); Atrial Tachycardia; Typical Atrial Flutter; Paroxysmal Atrial Fibrillation (PAF)
MeSH Terms: conditions — Tachycardia, Ventricular; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, single-arm, non-randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients of complex arrhythmias treated with EasyStars™ High Density Mapping Catheter (Experimental)
  Interventions: Device: EasyStars™ High Density Mapping Catheter

INTERVENTIONS:
Device: EasyStars™ High Density Mapping Catheter — All patients underwent treatment for complex arrhythmias using EasyStars™ High Density Mapping Catheter.

SUMMARY:
The primary objective of this study was to evaluate the clinical feasibility, safety, and surgical characteristics of the EasyStars™ High Density Mapping Catheterin in patients with complex arrhythmias.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the clinical feasibility, safety, and surgical characteristics of the EasyStars™ High Density Mapping Catheterin in patients with complex arrhythmias. In addition, the study assessed the catheter's usability and mapping performance through postoperative physician feedback.

ELIGIBILITY:
1. Clinical diagnosis: Ventricular tachycardia (VT)

   * Inclusion criteria:

     1. Patients aged between 18 and 80 years;
     2. Confirmed diagnosis of ventricular tachycardia (VT) via electrocardiogram (ECG) or 24-hour Holter monitoring;
     3. The patient has experienced at least one episode of VT in the past 6 months and exhibits symptoms of sustained or paroxysmal ventricular tachycardia;
     4. The patient meets the criteria for ablation surgery and has clear indications for ablation;
     5. The patient is in good general health and able to tolerate surgery (no severe underlying heart disease, such as severe heart failure or severe coronary artery disease);
     6. Voluntarily participates and signs an informed consent form.
   * Exclusion criteria:

     1. Uncontrolled heart failure (New York Heart Association functional class III-IV);
     2. History of acute or progressive myocardial infarction;
     3. Severe pulmonary, hepatic, or renal disease;
     4. Valvular heart disease or congenital heart disease;
     5. Excessive use of medications or medication intolerance (e.g., beta-blockers, antiarrhythmic drugs);
2. Clinical diagnosis: Atrial tachycardia (AT)

   * Inclusion criteria:

     1. Patients aged 18 to 80 years;
     2. Diagnosed with atrial tachycardia (AT) by electrocardiogram (ECG) or Holter monitoring;
     3. Patients presenting with clinical symptoms such as palpitations, chest tightness, or fatigue;
     4. Patients diagnosed with persistent or paroxysmal atrial tachycardia and meeting the criteria for ablation therapy;
     5. Patients who voluntarily participate and sign an informed consent form.
   * Exclusion criteria:

     1. Patients with severe valvular heart disease or congenital heart disease;
     2. Patients with severe left ventricular or right ventricular heart failure;
     3. Patients with severe systemic diseases, such as liver failure, kidney failure, or tumours;
     4. Patients with cardiomyopathy or aortic dissection;
3. Clinical diagnosis: atypical atrial flutter (AFL)

   * Inclusion criteria:

     1. Patients aged 18 to 80 years;
     2. Patients diagnosed with atypical atrial flutter (AFL) via electrocardiogram (ECG) or Holter monitoring;
     3. Patients with clinical symptoms (e.g., palpitations, chest tightness, fatigue, etc.) that significantly impair their quality of life;
     4. Patients who meet the criteria for atrial tachycardia ablation and have no other severe comorbidities;
     5. Voluntarily participate and sign an informed consent form.
   * Exclusion criteria:

     1. Patients with severe heart disease, such as cardiomyopathy or severe valvular disease;
     2. Patients with severe pulmonary disease, such as pulmonary arterial hypertension;
     3. Patients with a history of major cardiac surgery (e.g., heart transplantation);
4. Clinically diagnosed with paroxysmal atrial fibrillation (PAF)

   * Inclusion criteria:

     1. Patients aged 18 to 80 years;
     2. Diagnosed with paroxysmal atrial fibrillation (PAF) via electrocardiogram (ECG) or Holter monitoring;
     3. Frequent episodes of paroxysmal atrial fibrillation with symptoms such as palpitations, fatigue, and dyspnoea, and meeting the criteria for ablation;
     4. No other severe cardiac or systemic diseases, and meeting the criteria for ablation;
     5. Voluntarily participating and signing the informed consent form.
   * Exclusion criteria:

     1. Patients with severe valvular heart disease, aortic dissection, or cardiomyopathy;
     2. High-risk patients with a history of anticoagulant therapy or currently receiving anticoagulant therapy (e.g., history of thrombosis or stroke);
     3. Patients with severe underlying conditions such as cancer or severe diabetes;
5. Clinical diagnosis: Persistent atrial fibrillation (PsAF)

   * Inclusion criteria:

     1. Patients aged 18 to 80 years;
     2. Diagnosed with persistent atrial fibrillation (PsAF) via electrocardiogram (ECG) or Holter monitoring;
     3. Atrial fibrillation persisting for more than 7 days and symptoms affecting the patient's quality of life;
     4. Clear indications for ablation and no other severe comorbidities;
     5. Voluntarily participating and signing an informed consent form.

Exclusion criteria:

1. Presence of severe valvular heart disease or cardiomyopathy;
2. History of stroke or clinical evidence of thrombus formation;
3. Severe heart failure (NYHA III-IV class);
4. High-risk cardiac conditions (e.g., acute myocardial infarction, coronary artery disease); In the above different types of rapid arrhythmias, the inclusion criteria primarily focus on the diagnosis and control of clinical symptoms for different types of arrhythmias, while the exclusion criteria focus on avoiding patients with severe comorbidities or those unable to tolerate surgery. Through this patient screening method, the safety of the study and the accuracy of the data are ensured, thereby enabling a better assessment of the clinical efficacy of the new EasyStars catheter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
primary efficacy endpoint | On the day of the surgery
  The proportion of immediate success (all participating subjects) in treating rapid arrhythmias using EasyStars™ High Density Mapping Catheter in combination with cardiac ablation catheters and three-dimensional cardiac electrophysiology mapping systems